CLINICAL TRIAL: NCT05267795
Title: Reducing Pain Thresholds Using a Focused Music Listening Technique
Brief Title: Reducing Pain With Focused Music Listening
Acronym: PainMusic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFS Toppforsk
Record Dates: First submitted 2022-01-31; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The experiment used a 2x2 within-subjects design in which participants either listened to music or underwent a silent control period and either performed an active foot tapping task, or a passive control task with no movement resulting in four experimental trial types: (a) Music Active (music with tapping); (b) Music Passive (music without tapping); (c) Silence Active (silence with tapping); and (d) Silence Passive (silence without tapping). The allocation of the music excerpts to the task (active, passive) was random, and the order of the four experimental trial types was counterbalanced. Specific pain levels were applied on the participants' fingernails in each of 40 experimental trials using pressure algometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operationalization (Experimental): The experiment used a 2x2 within-subjects design in which participants either listened to music or underwent a silent control period and either performed an active foot tapping task, or a passive control task with no movement resulting in four experimental trial types: (a) Music Active (music with tapping); (b) Music Passive (music without tapping); (c) Silence Active (silence with tapping); and (d) Silence Passive (silence without tapping). The allocation of the music excerpts to the task (active, passive) was random, and the order of the four experimental trial types was counterbalanced.
  Interventions: Behavioral: Experimentally-induced pain

INTERVENTIONS:
Behavioral: Experimentally-induced pain — Specific pain levels were applied on the participants' fingernails in each of 40 experimental trials using pressure algometry.

SUMMARY:
Pain-reducing effects of music listening are well-established, but the effects are small and their clinical relevance questionable. Recent theoretical advances, however, have proposed that synchronizing to music, such as clapping, tapping or dancing, has evolutionarily important social effects that are associated with activation of the endogenous opioid system (EOS; which supports both analgesia and social bonding). Thus, active sensorimotor synchronization to music could have stronger analgesic effects than simply listening to music. However, to the best of the investigators' knowledge, the hypothesis of an EOS activation by sensorimotor synchronization to music has never been investigated. Accordingly, the investigators set up a test with the premise that if sensorimotor synchronization to music indeed activates the EOS, then it should have larger pain-reducing effects than simply listening to music. Using pressure algometry to the fingernails, specific amounts of pain were delivered to healthy adults either during music listening or silence, while either performing an active tapping task or a passive control task. As the dependent variable, perceived pain was rated on a scale ranging from 1 to 9 (1 = very little, 5 = medium, 9 = very strong). In addition, to pain ratings, participants provided ratings of their emotional state in terms of pleasantness as well as arousal, and then rated their familiarity with the music (also on scales ranging from 1 to 9). Emotion ratings were obtained to explore whether the mechanisms driving pain-reducing effects of sensorimotor synchronization to music include emotion. At the end of the experiment, participants also rated their preference for the music on a scale ranging from 1 to 9 (see Method). Familiarity and preference ratings were obtained to elucidate possible contributions of these factors on pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Healthy

Exclusion Criteria:

* History of a psychiatric or neurological disease
* History of substance dependence
* use of any prescription drugs
* Hearing impairment
* Musical anhedonia

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Perceived Pain | 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very little, 5 = medium, 9 = very strong)
Emotional state with regard to felt pleasantness | 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very uncomfortable, 5 = medium, 9 = very comfortable)
Emotional state with regard to felt arousal | 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very calm, 5 = medium, 9 = very activated)
Familiarity with the music excerpt (only during trials with music) | 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = not at all, 5 = partially known, 9 = well known)
Preference ratings for each musical excerpt | 5 min (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = strongly disliked, 5 = medium, 9 = strongly liked)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Koelsch, PhD, Principal Investigator — University of Bergen, Norway
Locations (1):
- University of Bergen, Bergen, Bergen Municipality, Norway

REFERENCES:
- [Derived] Werner LM, Skouras S, Bechtold L, Pallesen S, Koelsch S. Sensorimotor synchronization to music reduces pain. PLoS One. 2023 Jul 28;18(7):e0289302. doi: 10.1371/journal.pone.0289302. eCollection 2023. PMID 37506059